CLINICAL TRIAL: NCT04406974
Title: Locally Advanced Colorectal Cancer and Recurrence After Colorectal Cancer in Region Västra Götaland
Brief Title: Locally Advanced Colorectal Cancer and Local Recurrences in Västra Götaland
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Eva Angenete, Professor, Sahlgrenska University Hospital
Other Study IDs: Lokalrecidiv i VGR
Record Dates: First submitted 2020-05-24; First posted 2020-05-29 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative; Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with local recurrence
  Interventions: Procedure: Surgery or treatment for local recurrence; Procedure: Surgery for advanced colorectal cancer
- Patients with advanced colorectal cancer
  Interventions: Procedure: Surgery or treatment for local recurrence; Procedure: Surgery for advanced colorectal cancer

INTERVENTIONS:
Procedure: Surgery or treatment for local recurrence — Surgery or treatment for local recurrence
Procedure: Surgery for advanced colorectal cancer — Surgery for advanced colorectal cancer

SUMMARY:
The aim of this study is to review the treatment strategies of locally advanced colorectal cancer and locally recurrent rectal cancer in Västra Götaland during 1995-2016. The aim is to evaluate time trends and outcome both related to morbidity and cancer specific survival, we will also evaluate the results after advanced reconstruction. The study will identify the population using the Swedish ColoRectal Cancer Registry and then the individual patient charts will be reviewed. The data will be collected in a clinical record form covering demography (age, sex, co-morbidity, BMI and diagnoses) as well as treatments strategy, surgical procedures, re-operations, complications, readmissions, hospital stay, stoma formation etc.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal cancer
* Local recurrence for colorectal cancer
* Curative treatment for colorectal cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in Region Västra Götaland 1995-2018 for colorectal cancer will be identified using the local Swedish Colorectal Cancer Registry. Further selection will depend on the primary outcome in substudies.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Survival after local recurrence | 3 years
Risk factors for local recurrence | Preoperative data, about 1 month prior surgery
Complications after urinary reconstruction surgery for locally advanced cancer | 90 days
Patient experiences after local recurrence | 3 years postopeartively after local recurrence
  Indepth interviews with patients with local recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Surgery, Sahlgrenska University Hospital/Ostra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided